CLINICAL TRIAL: NCT01597882
Title: Improved Targeting of Admission Avoidance Interventions in Older People With Long-term Conditions:An Observational,Longitudinal Study Exploring the Feasibility of Measures of Strength as a Monitoring Aid in Patients Receiving Case Management
Brief Title: Improving Monitoring of Patients Receiving Case Management
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Principal Investigator, Nicola Barnes, Post-graduate Research Student, University of Southampton
Other Study IDs: 8550; 1409-ERGO (Other: University of Southampton)
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Conditions; Coronary Heart Disease; Diabetes; Hypertension; Chronic Obstructive Pulmonary Disease
Keywords: case management; long term conditions; aged sixty five and over
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus; Hypertension; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Case managed patients: Patients aged 65 years and over receiving community case management.

SUMMARY:
The UK population is ageing and the likelihood of having a long term health condition increases with age. Three out of every five people over 60 in the UK have a long term condition. Ageing and having a long term condition increases the chance of having difficulty being independent and carrying out day to day activities. In recent years the NHS has made a greater effort to prevent these difficulties in patients with long term conditions.

One approach to help patients with long term conditions is case management, where by (usually) a community matron visits patients at home, looking for early warning signs of any worsening of their condition and arranging care and treatment. But the current way this is done varies across the country and hospital admissions are still rising. In order to give the right care at the right time, effective monitoring is needed to help the community matron detect and act on changes in the patient's condition.

Loss of muscle strength in old age is linked to a poor health, but it is not known whether simple measures of muscle strength could be used to detect and predict declines in health in the short to medium term to help maintain independence and prevent an accident or hospital admission.

The aim of this study is to look at whether monitoring muscle strength in case managed patients is practical, acceptable and useful in detecting when a patient's condition worsens. Each patient will be visited by the researcher in their home twice in the first week, then once every two weeks, for another 5 weeks, to carry out three simple measures of grip and respiratory strength, and complete questionnaires about their health and ability to carry out day to day activities. Each visit will last about 20 to 30 minutes. A small group of clinicians will be asked about their views of the strength measures. Database analysis will allow descriptive data on the patient group to be gathered and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or over receiving health case management in the community.

Exclusion Criteria:

1. Enrolled in any other research study
2. Preclude consent:

   * Significant cognitive impairment resulting in lack of capacity to consent. b. Unable to communicate without significant aids e.g. Non-English speaking.
3. Preclude participation/ collection of data

   * Significant emotional distress or psychotic illness active within the last 6 months.
   * Receiving end of life care.
   * Current illness that would preclude data collection.
   * Upper limb pathology that would limit participation e.g. bone fracture within the previous 6 months.
   * Identified as high risk patients with regards to lone working safety by their case manager.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients receiving cmmunity health case management.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Grip strength | 13 weeks
  To assess reliability of measure over a one week period and the stability of the measure over 13 weeks, in this patient group, as well as acceptability.

SECONDARY OUTCOMES:
Peak expiratory flow | 13 weeks
  To measure reliability over one week and stability over 13 weeks in this patient group, as well as acceptability.
Peak inspiratory flow | 13 weeks
  To assess reliability over one week, and stability over 13 weeks in this patient group, as well as acceptability.
Sickness behaviour scale | 13 weeks
  To explore the relationship between sickness behaviour and measures of strength.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Barnes, MPharm, Principal Investigator — University of Southampton
Locations (2):
- United Kingdom (2):
  - Solent NHS Trust, Portsmouth
  - Southern Health NHS Foundation Trust, Southampton